CLINICAL TRIAL: NCT03884816
Title: Longitudinal Incidence Study in Subtype B-Prevalent Region Among Men Who Have Sex With Men at Risk for Human Immunodeficiency Virus (HIV) Infection to Determine Feasibility of HIV Vaccine Efficacy Trials
Brief Title: HIV and STIs Clinical Study in Germany
Status: Completed | Type: Observational
Sponsor: Hendrik Streeck (Other)
Collaborators: US Military HIV Research Program (Network); United States Army Medical Materiel Development Activity (U.S. Federal Agency); Federal Ministry of Health, Germany (Other Government); German Center for Infection Research (Other)
Responsible Party: Sponsor-Investigator, Hendrik Streeck, Prof. Dr. med. Hendrik Streeck, University Hospital, Essen
Organization: University Hospital, Essen (Other)
Other Study IDs: BRAHMS Study
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: HIV Infections; Sexual Behavior; Risk Reduction
Keywords: HIV; Pre-exposure prophylaxis; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexual Behavior; Risk Reduction Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, blood (serum, plasma), swabs (oral, rectal)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determine the Incidence and Retention Rate — Determine the incidence of HIV and the retention rate of MSM/TGW/TGM/Intersex at risk for HIV infection

SUMMARY:
The BRAHMS study is a prospective observational cohort study aiming to investigate how often people that are at risk to get infected with HIV contract HIV and how long people stay in the study. The University Hospital Essen is interested in finding out how often participants contact other sexually transmitted infections (STI) and hepatitis as well as in the development of HIV vaccines to test in the future. The University Hospital Essen will therefore also ask participants to fill out a questionnaire asking their general willingness to participate in such a trial (i.e., where the vaccine might be targeted to an HIV subtype not as common in Europe) to understand whether such testing would be possible in the future in Germany.

DETAILED DESCRIPTION:
In Germany, new HIV diagnoses are steadily increasing again since 2000. 74% of infected individuals living in Germany are men who have sex with men (MSM) whereas only 15% were infected by heterosexual contact. The HIV epidemic is mainly restricted to big cities such as Cologne, Berlin, Hamburg. The successful conduct of HIV vaccine efficacy trials requires recruitment, enrolment, and long-term retention of informed, willing, and HIV-negative but at-risk participants. Therefore, the University Hospital Essen plans a vaccine preparedness study to assess the feasibility of future HIV vaccine efficacy trials in Germany, a subtype B prevalent region in Europe, as this has never been assessed in Germany.

Notably investigators conduct a cohort study to characterize HIV incidence and retention among high risk, HIV uninfected MSM/Transgender women (TGW)/Transgender Men (TGM)/Intersex in the setting of prevention modalities that may be available to participants, including PrEP and regular HIV risk reduction counselling and testing. The design of the study will address several unique questions about the community at highest risk for HIV infection and will provide strong data for prevention methods including PrEP.

Moreover, it has been clearly demonstrated that sexually transmitted infections (STIs) can increase the risk of acquiring a HIV infection. Therefore, early diagnosis and treatment of STI is crucial to reduce this risk factor of HIV acquisition and to inform individuals about their risk to become HIV infected. As STIs are a crucial factor in the scope of an incidence analysis of HIV in MSM and are underdiagnosed often, extensive screening measures are implemented within the study to an extent never performed in Germany before.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-uninfected
2. 18-55 years of age
3. Male sex - (at birth, chosen or intersexual)
4. Able and willing to give informed consent
5. Able to read and write in German or English language
6. Willing to provide identification card
7. Willing to be followed for 12 months in the study and undergo study procedures including testing for HIV and receipt of HIV test results
8. Willing to provide contact information for themselves and, if available, one personal contact who would know their whereabouts during the study period
9. Willing to provide information regarding risk behaviors
10. Demonstrates any one of the following risk factors:

    1. reports condomless anal intercourse with at least two unique male partners in the past 24 weeks (partners must be either HIV-infected or of unknown HIV status) or
    2. documented history (lab work, physician's note etc.) of syphilis in the past 24 weeks or
    3. documented history of rectal gonorrhea or chlamydia in the past 24 weeks or
    4. documented history of rectal mycoplasma genitalium in the past 24 weeks or
    5. documented history of acute Hepatitis C virus (HCV) infection in the past 24 weeks

Exclusion Criteria:

1. Any significant condition (including medical, psychologic/psychiatric and social) which, in the judgment of the study investigator, might interfere with the conduct of the study or be detrimental to the participant.
2. Participation in a previous HIV vaccine study, unless documented placebo recipient.
3. Concurrent participation in investigational agents for treatment or prevention of HIV-1 infection (e.g. Discover Study)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men who have sex with Men (MSM) Transgender Women (TGW) Transgender Men (TGM) Intersex
Study Population: The study population will consist of 1,000 HIV uninfected MSM/TGW/TGM/Intersex ages 18-55 years at risk for HIV infection at all study sites. Incidence rate will be evaluated across all sites as a primary objective. Each participant will be followed for a total of 12 months with assessment of HIV and STI status and risk behavior conducted at screening, three months (V2), six months (V3), nine months (V4), and twelve months (V5). It is anticipated that total accrual will take approximately 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Incidence of HIV in a cohort of MSM/TGW/TGM/Intersex at risk for HIV infection | Through study completion, an average of 2 years
  Descriptive statistics will be generated to summarize incidence (as measured as new HIV infections occurring during the study period) HIV infections. The power calculation targets a 3% incidence rate per year. An overall estimate of HIV incidence and 95% confidence intervals (CI) will be estimated assuming a Poisson distribution.
Retention rate of MSM/TGW/TGM/Intersex at risk for HIV infection in a cohort study | Through study completion, an average of 2 years
  The primary assessment of retention will be conducted assuming a binomial distribution and individuals will be considered retained at 12 months if they complete the final study visit. Retention will also be estimated with a 95% CI for each study visit. Factors associated with overall retention will be assessed in a logistic regression model.

SECONDARY OUTCOMES:
Prevalence of HIV infection among screened participants | At screening (until last participant in), an average of 1 year
  Descriptive statistics will be generated to summarize prevalence (as measured as HIV positive cases study period) HIV infections. Once enrolment is completed, baseline HIV prevalence will be calculated.
Relationship between certain behavior and risk of HIV infection | Through study completion, an average of 2 years
  Participants will receive questionnaires. The risks of HIV infection will be based on factors such as sexual behavior, pre- and post-exposure prophylaxys and others. Descriptive statistics will be generating to summarize risk factors associated with HIV infection.
Willingness of MSM/TGW/TGM/Intersex at risk for HIV infection to participate in a future HIV vaccine trial | At visit 1 and 5 (visit 1 is day 0, visit 5 is day 364)
  Willingness to participate in an HIV vaccine trial will be estimated assuming a binomial distribution. Factors associated with willingness to participate in vaccine trial will be evaluated using logistic regression models.
Prevalence of STIs in MSM/TGW/TGM/Intersex at risk for HIV infection | At screening (until last participant in), an average of 1 year
  Descriptive statistics will be generated to summarize prevalence (as measured as STIs positive cases study period) STI infections. Once enrolment is completed, baseline STI prevalence will be calculated.
Incidence of STIs in MSM/TGW/TGM/Intersex at risk for HIV infection | Through study completion, an average of 2 years
  Descriptive statistics will be generated to summarize incidence (as measured as new STI infections occurring during the study period) STI infections. An overall estimate of STI incidence and 95% confidence intervals will be estimated assuming a Poisson distribution.
Attitudes regarding pre-exposure prophylaxis (PrEP) among MSM/TGW/TGM/Intersex at risk for HIV infection | At screening and at visit 1,2,3,4 and 5 (visit 1 is day 0, visit 2 is day 84, visit 3 is day 168, visit 4 is day 252, visit 5 is day 364)
  Attitudes regarding PrEP will be evaluated using questionnaires. Behavioural questionnaire over time will be assessed by frequency tables and bar graphs.
Relative HIV incidence between MSM/ TGW/TGM/Intersex across sites | Through study completion, an average of 2 years
  Descriptive statistics will be generated to summarize incidence (as measured as new HIV infections occurring during the study period) HIV infections. The power calculation targets a 3% incidence rate per year. Data may be compared across sites for comparison and evaluation of factors impacting incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Streeck, Prof. Dr., Principal Investigator — Institute for HIV Research
Locations (10):
- Germany (10):
  - Praxis Dr. Cordes, Berlin
  - Zentrum für Infektiologie Berlin Prenzlauer Berg (ZIBP), Berlin
  - Praxis Jessen, Berlin
  - WIR "Walk In Ruhr", Bochum
  - Praxis Hohenstaufenring, Cologne
  - Universitätsklinikum, Cologne
  - HPSTD clinic, Essen
  - Infektiologikum, Frankfurt am Main
  - ifi-Institut für interdisziplinäre Medizin, Hamburg
  - Interdisziplinäres HIV-Zentrum am Klinikum rechts der Isar (IZAR), München

IPD SHARING:
Plan to Share IPD: Yes
The study collaborators recognize the importance of disseminating scientific and medical study data as soon as the study data sets are complete and analyzed; therefore, the study leadership would encourage their presentation, discussion and publication at seminars or conferences (national, regional and international) and in reputable scientific journals in open access. All publications resulting from this study will be cleared through the collaborating partners to the study. Anonymous data can be obtained upon request to the PI of the study. Confidentiality of participants will be maintained by the fact that no individual results will be reported or published, only group/aggregate results. Data collected during the trials that underlie the results presented in scientific publications will be shared. Distribution of study data must be always approved by the scientific steering committee of the study and final approval needs to be obtained by the PI.
Time Frame: After publication. No end date
Access Criteria: Researchers who would like to access the data after completion of trial should provide a written request to studien@hiv-forschung.de

REFERENCES:
- See also: Study Information (see cohort studies BRAHMS Study) — http://www.hiv-forschung.de